CLINICAL TRIAL: NCT05014269
Title: Phacoemulsification in Patients With Corneal Opacities Using Slit Illumination of the Surgical Microscope
Brief Title: Phacoemulsification in Patients With Corneal Opacities
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud F. Rateb, Assistant professor of Ophthalmology, Assiut University
Other Study IDs: phacoemulsification surgery
Record Dates: First submitted 2021-08-09; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Senile Cataract
Keywords: Senile Cataract; Corneal opacity; Phacoemulsification
MeSH Terms: conditions — Corneal Opacity | interventions — Phacoemulsification; Vision, Ocular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Phacoemulsification in eyes with corneal opacities — senile cataract extraction using lens emulsification under the slit illuimnation of the surgical microscope

SUMMARY:
In this retrospective case series, the feasibility of performing phacoemulsification using slit illumination in eyes with corneal opacity was assessed.

DETAILED DESCRIPTION:
Corneal opacity is often encountered in patients seeking senile cataract surgery in developing countries. Corneal opacity impairs the intraoperative visualization during cataract surgery which increases the risk of copmlications.

Several techniques were described to enhance the intraoperative visualization such as the use of anterior endoscopy, chandeiler retroillumination, and anterior chamber endoillumination. All these techniques require costly instrumentation.

the aim of this study was to assess the feasibility of performing phacoemulsification using slit illumination of the surgical microscope without the need of additional instruments, and report the visual outcome.

ELIGIBILITY:
Inclusion criteria:

* The presence of visually significant senile cataract.
* A recent history of progressive diminution of vision within few months.
* Stable density and size of a preexisting trachomatous corneal opacity that does not impair the pupil or lens visualization after pupillary dilatation.

Exclusion Criteria:

* History of trauma, infectious corneal ulcers, or intraocular surgery.
* Coexisting ocular diseases e.g. glaucoma, retinal detachment, and vitreous hemorrhage.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with visually significant senile cataract and corneal opacities
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The rate of intra-operative complications of phacoemulsification in eyes with corneal opacities using the slit ilumination of the surgical microscope. | 3 months
  the frequency of the intraoperative complications of phacoemulsification in eyes with corneal opacities

SECONDARY OUTCOMES:
Visual outcome of phacoemulsification in eyes with corneal opacities | 3 months
  meaurement of the change of the distance corrected visual acuity bafoer after phacoemulsification using Snellen chart